CLINICAL TRIAL: NCT06931795
Title: Implementation of a HABIT-ILE Intervention at the William Lennox Neurological Centre for Sub-acute Adult Post-stroke Patients (<6 Mois): a Randomised Controlled Trial
Brief Title: Implementation of a HABIT-ILE Intervention at William Lennox Neurological Hospital (NeuREHA) - Adult
Acronym: Ad-NeuREHA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Université Catholique de Louvain (Other)
Responsible Party: Principal Investigator, Yannick Bleyenheuft, Professor, Université Catholique de Louvain
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B0392023000045
Record Dates: First submitted 2025-04-09; First posted 2025-04-17 (Actual); Last update posted 2025-04-17 (Actual); Status verified 2025-04

CONDITIONS: Stroke
Keywords: stroke, intensive intervention, motor skill learning, subacute
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HABIT-ILE (Experimental): Hand and arm bimanual intensive therapy including lower extremities
  Interventions: Behavioral: HABIT-ILE
- Conventional Intervention (Active Comparator): Conventional physical and occupational therapy (same amout of hours)
  Interventions: Behavioral: Conventional intervention

INTERVENTIONS:
Behavioral: HABIT-ILE — 2 weeks HABIT-ILE
  Other Names: HABIT-ILE Stroke
  Arms: HABIT-ILE
Behavioral: Conventional intervention — 2 weeks usual intervention (waitlist group)
  Arms: Conventional Intervention

SUMMARY:
Using a randomized controlled trial design, in an hospital environment, possible changes induced by the "Hand-arm Bimanual Intensive Therapy Including Lower Extremities (HABIT-ILE)" treatment program will be investigated in functional activities of daily living, motor and cognitive assessment of patients with sub-acute post-stroke

DETAILED DESCRIPTION:
The aim is to investigate, for the first time, the effectiveness of HABIT-ILE therapy in a hospital setting in the treatment of a population representative of the clinical population for adult patients with subacute stroke.

The hypothesis is that an in-hospital HABIT-ILE protocol will be more effective than conventional therapies usually given to patients with sub-acute post-stroke, and that this difference will be objectively demonstrated by clinical assessments of motor function, cognition and participation conducted before and after treatment periods.

The aim of the study is therefore to evaluate the effect of intensive bimanual hand-arm therapy including the lower extremities (HABIT-ILE) on body functions and structures, activity and participation in adulte patients suffering from subacute stroke..

ELIGIBILITY:
Inclusion Criteria:

* Phase aiguë ou subaiguë

Exclusion Criteria:

* Epilepsie instable
* Absence à déterminer sa volonté à participer
* Traitement toxine pendant le stage

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-04-15 (Estimated); Primary Completion 2026-12-20 (Estimated); Study Completion 2026-12-24 (Estimated)

PRIMARY OUTCOMES:
Changes on the Adult Assisting Hand Assessment Stroke (Ad-AHA Stroke) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  This assessment is an observation-based instrument assessing the effectiveness of the spontaneous use of the affected hand when performing bimanual activities in adults post stroke scored in a logit based 0-100 AHA-unit scale (higher score indicate higher ability)

SECONDARY OUTCOMES:
Changes in upper extremities sensorimotor functions assess by the Fugl-Meyer Assessment (FMA-UE) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The FMA-UE assess reflex activity, movement control and muscle strength in the upper extremity of people with post-stroke hemiplegia. Maximum score is 66 points (Higher scores indicates better functioning levels)
Changes in unimanual dexterity: Box and Blocks test (BBT) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The BBT is a test of gross manual dexterity. Each hand is tested individually and the BBT is scored through the number of blocks carried over the partition from one part to another part of a box during the one-minute trial period.
Changes in Canadian Occupational Performance Measure (COPM) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  This is an interview-setting designed to capture a patient's self-perception of performance and satisfaction of it in everyday activities, observed over time. During the interview, parents set up 5 activities considered difficult in daily life. These are then assessed, in a 1 to 10 scale, regarding the child's self-perception of performance and satisfaction of it. The total score is the average of the scores for perception and satisfaction separately (score from 1 to 10; higher score means better performance/satisfaction)
Changes in the Stroke Impact Scale (SIS) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  Self-reported questionnaire assessing multidimensional repercussions of the Stroke (strength, hand function, daily life activities, mobility, communication, emotion, memory, thinking and participation). Domains are scored on a metric of 0 to 100 (higher scores indicate better self-reported health)
Changes in activities of daily living assessed by ACTIVLIM-Stroke Questionnaire | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The ACTIVLIM-Stroke questionnaire measures a patient's ability to perform daily activities requiring the use of the upper and/or lower extremities through 20 items specific to patients after stroke. It ranges from - 6 to +6 logits (higher score means better performance).
Changes in activities of daily living assessed by ABILHAND Questionnaire | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The ABILHAND questionnaire specific to patients with chronic stroke measures a patient's manual ability to manage daily activities that require the use of the upper extremities, whatever the strategies involved, through 23 items. It ranges from -6 to +6 logits (higher score means better performance).
Changes in visual neglect assessed by the Bells Test | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The Bells Test is a cancellation test that allows for a quantitative and qualitative assessment of visual neglect in the near extra personal space. The patient score is based on the amount of time they take to complete the task, and the number of correct items (35 bells) they identify.
Changes in the Montreal Cognitive Assessment (MoCA) test | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The MoCA is a brief screening instrument originally designed to identify mild cognitive impairments in elderly patients attending a memory clinic. MoCA evaluates different domains (visuospatial abilities, executive functions, short-term memory recall, attention, concentration, working memory, language, and orientation to time and space) having a total of 30 points (higher scores indicate better self-reported health)
Changes in balance control assessed by the mini Balance Evaluation System Test (mini BEST test) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The miniBEST test is a shortened version of the Balance Evaluation Systems Test (BESTest). It assesses 6 different balance control systems, the BESTest was shortened based on factor analysis to include dynamic balance only (Higher scores indicate better performance). The test is a 14-item test scord on a 3-level ordinal scale (0-2). higher score means better performance.
Changes in the Two Minutes' Walk Test (2MWT) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The 2MWT assess endurance while walking 2 minutes without pause. More distance walked (in meters) indicate better performance.
Changes in National Institutes of Health Stroke Scale (NIHSS) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The National Institutes of Health Stroke Scale (NIHSS) is a 15-item impairment assessment scale designed to evaluate the neurological consequences and degree of recovery of a stroke patient. The scale assesses level of consciousness, extraocular movements, field of vision, facial muscle function, strength of extremities, sensory function, coordination (ataxia), language (aphasia), speech (dysarthria) and hemineglect (neglect).
Changes in Tardieu Scale et Modified Tardieu Scale (MTS) | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)
  The Tardieu Scale and Modified Tardieu Scale (MTS) are clinical measures of muscle spasticity for use in patients with neurological disorders. In the Tardieu Scale or the MTS, spasticity is quantified by assessing the response of the muscle when it is stretched at various velocities.
Changes in EQ-5D-5L | [Time Frame: T0 (baseline), T1 (after 2weeks intervention), T2(3 months follow-up)]
  The system comprises five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Each dimension has 5 levels: no problems, slight problems, moderate problems, severe problems and extreme problems. The patient is asked to indicate his/her health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state.

CONTACTS AND LOCATIONS:
Overall Officials: Yannick Bleyenheuft, PT, PhD, Professor, Principal Investigator — Insititue of Neurosciences, UCLouvain
Locations (2):
- Belgium (2):
  - Institute of Neurosciences, UCLouvain, Brussels
  - Spontaneous contact via doctors or other partners, Brussels

IPD SHARING:
Plan to Share IPD: No